CLINICAL TRIAL: NCT04011072
Title: Effect of Far Infrared Therapy on Arteriovenous Fistulas Maturation, Survival and Stenosis. A Randomized, Controlled Open-labeled Multicenter Study
Brief Title: Far Infrared Therapy on Arteriovenous Fistulas in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Hillerod Hospital, Denmark (Other); Holbaek Sygehus (Other); Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Kristine Lindhard, Principal Investigator, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIR HD
Record Dates: First submitted 2019-06-27; First posted 2019-07-08 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Arterio-venous Fistula
Keywords: Hemodialysis; Infrared therapy; Stenosis; Maturation; Arteriovenous fistula survival
MeSH Terms: conditions — Arteriovenous Fistula; Constriction, Pathologic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infrared treatment arm (Active Comparator): Far infrared radiation will be given for 40 minutes on the skin above the patients fistula in each dialysis session for one year
  Interventions: Radiation: Far infrared radiation
- Control arm (No Intervention): The control group will not receive any intervention, but will be followed with the same data as the treatment group

INTERVENTIONS:
Radiation: Far infrared radiation — The treatment group will receive FIR for 40 minutes on the skin above the fistula during each dialysis session for one year.
  Other Names: FIR
  Arms: Infrared treatment arm

SUMMARY:
The number of hemodialysis patients in the world are increasing. In order to receive a sufficient dialysis, the patients needs a well functioning and stable vascular access - preferably an arteriovenous fistula (AVF). Unfortunately, the AVF has a high incidence of stenosis with percutaneous trans luminal angioplasty (PTA) as the only treatment option and a short lifetime. Little do we know of how to improve the survival of the AVF.

With this study we want to explore the effect of far infrared therapy on the stenosis, maturation and survival of the arteriovenous fistula.

The investigators will divide the patients into 2 groups: A treatment group and a control group.

The treatment group will receive infrared therapy on their fistula during their dialysis session. The control group will not receive any infrared therapy.

The investigators hope to reduce the risk of stenosis in the fistula and improve the fistula survival with this treatment.

Furthermore, the investigators want to explore the change in several biochemical markers during the treatment with infrared therapy.

DETAILED DESCRIPTION:
Background:

The number of hemodialysis patients in the world are increasing. In order to receive an efficient dialysis, the patient needs a well-functioning and stable vascular access. Presently there is three options: an arteriovenous fistula (AVF), an arteriovenous graft (AVG) and a central venous catheter (CVC). CVCs are associated with an increased risk of stenosis of the central vessels, thrombosis in the AVF, infections and death. AVGs are associated with increased risk of infections, stenosis in the AVG and loss of access. This is why, the AVF is the preferred vascular access. But this vascular access does not come without risks. After the creation of an AVF there is a risk of 50 % for never maturing, which means the AVF cannot be used. Furthermore, the risk of stenosis in the AVF is also high, up to 67 % of the AVFs will have a stenosis, that needs an intervention. During this time the patient needs an alternative vascular access, such as a central venous catheter, which is related to an increased risk of infection, more hospital days and death.

The maturation of the AVF depends on several patient related, but also surgically related factors. Factors such as comorbidity, female sex, length of end stage renal disease, anatomy of the vessel, surveillance after AVF placement and the operations itself have all been shown to affect the AVF maturation. Fistula stenosis emerges from an endothelial dysfunction, inflammation and smooth muscle cell proliferation leading to intimal hyperplasia and in the end stenosis. Factors such as increased blood flow, inflammation, uremia and percutaneous transluminal angioplasty has been shown to affect the stenosis, It is not well understood, which molecular mechanism are responsible for the intimal hyperplasia.

There are few and not well established studies on how to improve the AVF survival and maturation.

Far infrared radiation (FIR) is an electromagnetic radiation (heat therapy), that is given directly on the skin above the AVF. In a few single center studies in Taiwan it has been shown to decrease the risk of stenosis and increase the fistula survival and maturation. However another study is disputing this. The mechanism behind FIR and better fistula survival is not fully understood. The infrared light is supposed to have a thermal effect, which leads to vasodilatation and a non-thermal effect, which influence the endothelial function and vasodilation and thereby it may decrease the inflammation and proliferation in the fistula, primarily through the releasing of several anti-inflammatory and vasodilating factors. This is not well documented.

Hypothesis:

Treatment with FIR for 40 minutes three times a week on the patients AVF will improve the AVF survival and maturation

Method:

This study is a randomized, controlled multicenter study on western patients

There will be 2 patient categories:

1. A group (82 patients) of dialysis patients with a newly created AF
2. A group (104 patients) of dialysis patients with an existing AVF

The patients will randomly be randomized 1:1 to either the treatment group or a control group. For group 2 the patients will be block randomized according to their access flow (AF) (above or below 950 ml/min). Furthermore these patients will be stratified according to interventions in there AVF (no interventions >/= 1 intervention) For the FIR treatment Ws Far Infrared Therapy Unit, model TY-102F (Medical device Class 11a CE0434) is being used. The patients will receive 40 minutes of infrared radiation on the skin of their fistula during each dialysis treatment for one year. The control group will not receive any FIR treatment, but will be followed according to the protocol and in line with the treatment group.

The patients will be followed until end of study or lost-to-follow-up (death, transplantations, change of renal replacement therapy, abandoned AVF, change of vascular access to CVC, consent withdrawal or if the patients moves away).

In order to explore the long term effects of FIR the patients will be followed for an extra 6 months according to the endpoints. In a subset of 2x20 patients of the randomized controlled trial we further wish to explore the influence of infrared therapy on endothelial function and inflammation during a FIR treatment session. Blood samples will be collected before and immediately after infrared treatment directly from the treatment site, since 2 needles are placed in the fistula during the dialysis treatment. The same samples will be collected in the control group and in the intervention group during the dialysis before the first infrared intervention in order to reduce the interindividual variation in the biomarkers.The changes in markers of endothelial dysfunction and inflammation during treatment and control dialysis session will be examined and compared.

Furthermore a blood sample from each patient will be collected at study start. The predictive value of the biomarkers of endothelial dysfunction and inflammation for the treatment response to infrared therapy and the prognosis for fistula maturation, stenosis and survival will be evaluated after the randomised controlled trial has ended.

Arterial stiffness (measured by Mobil-O-Graph) will also be evaluated as a marker for fistula survival and maturation.

A total of 186 participants will be recruited from 9 dialysis centres. If the study shows positive results, the implication of FIR in the clinic will have a huge beneficial effect for the hemodialysis patients vascular access and perhaps also patient survival. FIR is an easy treatment with a low cost-effectiveness and minimal or no side effects for the patient.

ELIGIBILITY:
Inclusion Criteria:

For incident AVF:

* Patients of 18 years of age or above
* Patients on chronic hemodialysis with a central venous catheter, who is having an AVF placed
* An AVF, that are maximum 3 weeks old

For prevalent AVF:

* Patients in chronic hemodialysis with a functioning AVF
* Patients of 18 yeas of age or above

Exclusion Criteria:

* Not obtainable informed consent
* Non compliant patients
* Patients who use both a CVC and an AVF as their vascular access
* Patient on both hemodialysis and peritoneal dialysis
* Planned living donor kidney transplantation
* Short life expectancy, less than a 1 year
* Patients on hemodialysis less than 3 times per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Time to fistula maturation for the incident fistulae | After 12 months
  Time from placement of the fistula to successful cannulation with 2 needles and successful hemodialysis treatment
Difference in number of fistula intervention for the prevalent fistulae | After 12 months
  For the fistulae with or without previous interventions we expect to find a decrease in the number of interventions in the treatment group compared to the control group

SECONDARY OUTCOMES:
Difference in number of fistula interventions in the incident fistula group | After 12 months
  Difference in the number of fistula intervention in the groups with a newly places fistula
Difference in the fistula diameter in the incident fistula group | After 12 months
  Is there a difference in the diameter measured by ultrasound between the 2 groups with patients with a newly places fistula
Number of abandoned fistulae in incident and prevalent groups | After 12 months
  For patients with a new fistula and patients with a fistula with/without interventions how many will loose their fistula and receive a new vascular access
The incidence of primary patency in the incident group | After 12 months
  How many of the fistulas in the group with a new fistula needs an intervention in order to get a functioning fistula
Number of patients with a never functioning fistula in the incident group | After 12 months
  How many patients in the newly places fistula group will never have a functioning fistula
Change in access flow in the incident and prevalent group | After 12 moths
  Does the access flow change between the control and treatment group
Baseline value in serum amyloid A as a predictor for AVF survival and stenosis | After 12 months
  Before study start the following markers will be explored : Serum Amyloid A (in Ug/ml),
Baseline value in adhesion molecules, heme-oxygenase and ADMA and selectin as a predictor for AVF survival stenosis | After 12 months
  Before study start the following change in markers will be explored: vascular cell adhesion molecule (in ng/ml), intercellular adhesion molecule (in ng/ml), sE-selectin (in ng/ml), assymetric dimethylarginine (in ng/ml), heme-oxygenase-1 (in ng/ml)
Baseline value in von willebrand factor as a predictor for AVF survival stenosis | After 12 months
  Before study start the following change in markers will be explored: vWF in ml-1)
Baseline in nitrite and nitrate as a predictor for AVF survival stenosis | After 12 months
  Before study start the following change in markers will be explored: nitrite (in uM), nitrate (in uM)
Baseline in different biomarkers as a predictor for AVF survival stenosis | After 12 months
  Before study start the following change in markers will be explored: endothelin (in pg/ml), prostaglandin E2 (in pg/ml, Interleukin-beta (pg/ml), Interleukin-6 (in pg/ml), Interleukin-8 (in pg/ml), tumor necrosis factor-alpha (in pg/ml), transformin growth factor-beta (in pg/ml) and monocyte chemoattractant protein 1 (in pg/ml).

OTHER OUTCOMES:
Difference in cannulation pain in the incident and prevalent group compared with visual analogue scale | After 12 months
  Do the patients receiving FIR treatment experience less pain during cannulation compared to the control group evaluated by the VAS (visual analogue scale) score
Difference in number with steal symptoms in the incident and prevalent group | After 12 months
  Is there a difference in patients with steal symptoms in the two groups
Acute changes in serum amyloid A after a single FIR treatment | After 40 minutes of FIR treatment
  In a subgroup of patients we want to study the acute changes of the following markers during a FIR treatment Analysing Serum Amyloid A (in Ug/ml)
Acute changes in adhesion molecules, heme-oxygenase and ADMA and selectin as a predictor for AVF survival stenosis after a single FIR treatment | After 40 minutes of FIR treatment
  In a subgroup of patients we want to study the acute changes of the following markers during a FIR treatment, analysing: vascular cell adhesion molecule (in ng/ml), intercellular adhesion molecule (in ng/ml), sE-selectin (in ng/ml), assymetric dimethylarginine (in ng/ml), heme-oxygenase-1 (in ng/ml)
Acute changes in von willebrand factor after a single FIR treatment | After 40 minutes of FIR treatment
  In a subgroup of patients we want to study the acute changes of the following markers during a FIR treatment Analysing: von WillebrandFactor (in ml-1)
Acute changes in nitrite and nitrate after a single FIR treatment | After 40 minutes of FIR treatment
  In a subgroup of patients we want to study the acute changes of the following markers during a FIR treatment Analysing: nitrite (in uM), nitrate (in uM)
Acute changes in different biomarkers after a single FIR treatment | After 40 minutes of FIR treatment
  In a subgroup of patients we want to study the acute changes of the following markers during a FIR treatment Analysing: endothelin (in pg/ml), prostaglandin E2 (in pg/ml), Interleukin-beta (pg/ml), Interleukin-6 (in pg/ml), Interleukin-8 (in pg/ml), tumor necrosis factor-alpha (in pg/ml), transformin growth factor-beta (in pg/ml) and monocyte chemoattractant protein 1 (in pg/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Ditte Hansen, Doctor, Study Chair — Herlev Hospital, Department of Nephrology
Locations (9):
- Denmark (9):
  - Rigshospitalet, Copenhagen
  - Frederiksberg Hospital, Frederiksberg
  - Herlev Hospital, Herlev
  - Hilleroed Hospital, Hillerød
  - Holbæk Hospital, Holbæk
  - Hvidovre Hospital, Hvidovre
  - Nykøbing Falster Hospital, Nykøbing Falster
  - Roskilde Hospital, Roskilde
  - Slagelse Hospital, Slagelse

REFERENCES:
- [Background] Lacson E Jr, Wang W, Hakim RM, Teng M, Lazarus JM. Associates of mortality and hospitalization in hemodialysis: potentially actionable laboratory variables and vascular access. Am J Kidney Dis. 2009 Jan;53(1):79-90. doi: 10.1053/j.ajkd.2008.07.031. Epub 2008 Oct 18. PMID 18930570
- [Background] Bray BD, Boyd J, Daly C, Donaldson K, Doyle A, Fox JG, Innes A, Khan I, Peel RK, Severn A, Shilliday I, Simpson K, Stewart GA, Traynor J, Metcalfe W; Scottish Renal Registry. Vascular access type and risk of mortality in a national prospective cohort of haemodialysis patients. QJM. 2012 Nov;105(11):1097-103. doi: 10.1093/qjmed/hcs143. Epub 2012 Aug 20. PMID 22908320
- [Background] Vascular Access Work Group. Clinical practice guidelines for vascular access. Am J Kidney Dis. 2006 Jul;48 Suppl 1:S248-73. doi: 10.1053/j.ajkd.2006.04.040. No abstract available. PMID 16813991
- [Background] Vanholder R, Canaud B, Fluck R, Jadoul M, Labriola L, Marti-Monros A, Tordoir J, Van Biesen W. Diagnosis, prevention and treatment of haemodialysis catheter-related bloodstream infections (CRBSI): a position statement of European Renal Best Practice (ERBP). NDT Plus. 2010 Jun;3(3):234-246. doi: 10.1093/ndtplus/sfq041. No abstract available. PMID 30792802
- [Background] Dhingra RK, Young EW, Hulbert-Shearon TE, Leavey SF, Port FK. Type of vascular access and mortality in U.S. hemodialysis patients. Kidney Int. 2001 Oct;60(4):1443-51. doi: 10.1046/j.1523-1755.2001.00947.x. PMID 11576358
- [Background] Rayner HC, Pisoni RL, Gillespie BW, Goodkin DA, Akiba T, Akizawa T, Saito A, Young EW, Port FK; Dialysis Outcomes and Practice Patterns Study. Creation, cannulation and survival of arteriovenous fistulae: data from the Dialysis Outcomes and Practice Patterns Study. Kidney Int. 2003 Jan;63(1):323-30. doi: 10.1046/j.1523-1755.2003.00724.x. PMID 12472799
- [Background] Al-Jaishi AA, Oliver MJ, Thomas SM, Lok CE, Zhang JC, Garg AX, Kosa SD, Quinn RR, Moist LM. Patency rates of the arteriovenous fistula for hemodialysis: a systematic review and meta-analysis. Am J Kidney Dis. 2014 Mar;63(3):464-78. doi: 10.1053/j.ajkd.2013.08.023. Epub 2013 Oct 30. PMID 24183112
- [Background] Smith GE, Gohil R, Chetter IC. Factors affecting the patency of arteriovenous fistulas for dialysis access. J Vasc Surg. 2012 Mar;55(3):849-55. doi: 10.1016/j.jvs.2011.07.095. Epub 2011 Nov 8. PMID 22070937
- [Background] Bashar K, Conlon PJ, Kheirelseid EA, Aherne T, Walsh SR, Leahy A. Arteriovenous fistula in dialysis patients: Factors implicated in early and late AVF maturation failure. Surgeon. 2016 Oct;14(5):294-300. doi: 10.1016/j.surge.2016.02.001. Epub 2016 Mar 15. PMID 26988630
- [Background] Brahmbhatt A, Remuzzi A, Franzoni M, Misra S. The molecular mechanisms of hemodialysis vascular access failure. Kidney Int. 2016 Feb;89(2):303-316. doi: 10.1016/j.kint.2015.12.019. PMID 26806833
- [Background] Lin CC, Liu XM, Peyton K, Wang H, Yang WC, Lin SJ, Durante W. Far infrared therapy inhibits vascular endothelial inflammation via the induction of heme oxygenase-1. Arterioscler Thromb Vasc Biol. 2008 Apr;28(4):739-45. doi: 10.1161/ATVBAHA.107.160085. Epub 2008 Jan 17. PMID 18202320
- [Background] Shui S, Wang X, Chiang JY, Zheng L. Far-infrared therapy for cardiovascular, autoimmune, and other chronic health problems: A systematic review. Exp Biol Med (Maywood). 2015 Oct;240(10):1257-65. doi: 10.1177/1535370215573391. Epub 2015 Feb 25. PMID 25716016 (Retraction: PMID 32686476 Exp Biol Med (Maywood). 2020 Aug;245(14):NP1)
- [Background] Lin CC, Yang WC, Chen MC, Liu WS, Yang CY, Lee PC. Effect of far infrared therapy on arteriovenous fistula maturation: an open-label randomized controlled trial. Am J Kidney Dis. 2013 Aug;62(2):304-11. doi: 10.1053/j.ajkd.2013.01.015. Epub 2013 Mar 6. PMID 23474008
- [Background] Lin CC, Chang CF, Lai MY, Chen TW, Lee PC, Yang WC. Far-infrared therapy: a novel treatment to improve access blood flow and unassisted patency of arteriovenous fistula in hemodialysis patients. J Am Soc Nephrol. 2007 Mar;18(3):985-92. doi: 10.1681/ASN.2006050534. Epub 2007 Jan 31. PMID 17267744
- [Background] Lai CC, Fang HC, Mar GY, Liou JC, Tseng CJ, Liu CP. Post-angioplasty far infrared radiation therapy improves 1-year angioplasty-free hemodialysis access patency of recurrent obstructive lesions. Eur J Vasc Endovasc Surg. 2013 Dec;46(6):726-32. doi: 10.1016/j.ejvs.2013.09.018. Epub 2013 Sep 25. PMID 24119468
- [Background] McGrogan DG, Stringer S, Cockwell P, Jesky M, Ferro C, Maxwell AP, Inston NG. Arterial stiffness alone does not explain arteriovenous fistula outcomes. J Vasc Access. 2018 Jan;19(1):63-68. doi: 10.5301/jva.5000791. PMID 29076519
- [Background] Dember LM, Imrey PB, Duess MA, Hamburg NM, Larive B, Radeva M, Himmelfarb J, Kraiss LW, Kusek JW, Roy-Chaudhury P, Terry CM, Vazquez MA, Vongpatanasin W, Beck GJ, Vita JA; Hemodialysis Fistula Maturation Study GroupFeldmanH.FarberA.KaufmanJ.SternL.LeSageP.KivorkC.SoaresD.MalikovaM.AllonM.YoungC.TaylorM.WoodardL.MangadiK.MundaR.LeeT.AllowayR.El-KhatibM.CanaanT.PflumA.ThiekenL.Campos-NaciffB.HuberT.BerceliS.JansenM.McCaslinG.TrahanY.DavidsonI.HwangC.LightfootT.LivingstonC.ValenciaA.DolmatchB.FenvesA.HawkinsN.CheungA.KinikiniD.TreimanG.IhnatD.SarfatiM.LavasaniI.MaloneyM.SchlotfeldtL.BuchananC.ClarkC.CrawfordC.HamlettJ.KundzinsJ.ManahanL.WiseJ.GassmanJ.GreeneT.LiL. Vascular Function at Baseline in the Hemodialysis Fistula Maturation Study. J Am Heart Assoc. 2016 Jul 22;5(7):e003227. doi: 10.1161/JAHA.116.003227. PMID 27451463
- [Background] Roy-Chaudhury P, Sukhatme VP, Cheung AK. Hemodialysis vascular access dysfunction: a cellular and molecular viewpoint. J Am Soc Nephrol. 2006 Apr;17(4):1112-27. doi: 10.1681/ASN.2005050615. PMID 16565259
- [Background] Lee T, Misra S. New Insights into Dialysis Vascular Access: Molecular Targets in Arteriovenous Fistula and Arteriovenous Graft Failure and Their Potential to Improve Vascular Access Outcomes. Clin J Am Soc Nephrol. 2016 Aug 8;11(8):1504-1512. doi: 10.2215/CJN.02030216. Epub 2016 Jul 11. PMID 27401527
- [Derived] Lindhard K, Hansen HP, Gliese K, Hansen E, Hommel K, Jensen B, Liem Y, Lindegaard-Pedersen B, Pourarsalan M, Rix M, Heaf J, Hansen D. The effect of far infrared radiation on maturation in arteriovenous fistulas in patients on hemodialysis: A randomized controlled, multicenter trial. J Vasc Access. 2025 Nov 3:11297298251385043. doi: 10.1177/11297298251385043. Online ahead of print. PMID 41178583
- [Derived] Lindhard K, Rix M, Heaf JG, Hansen HP, Pedersen BL, Jensen BL, Hansen D. Effect of far infrared therapy on arteriovenous fistula maturation, survival and stenosis in hemodialysis patients, a randomized, controlled clinical trial: the FAITH on fistula trial. BMC Nephrol. 2021 Aug 21;22(1):283. doi: 10.1186/s12882-021-02476-x. PMID 34419006